CLINICAL TRIAL: NCT02071407
Title: A Clinical Trial of the Effect of Midazolam on the Cerebral Metabolism and Inflammatory Response in Patients With Moderate and Severe Traumatic Brain Injury
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Subei People's Hospital of Jiangsu Province (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014021801
Record Dates: First submitted 2014-02-21; First posted 2014-02-25 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Traumatic Brain Injury
Keywords: traumatic brain injury; sedation; midazolam
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- N1(traditional treatment group) (Placebo Comparator): Patients in group N1 are treated with basic therapeutic measures which include reducing intracranial pressure with mannitol, hemostasis, acid inhibition, anti-infection, nutrition support and control of blood glucose, blood pressure and body temprature.
  Interventions: Drug: Placebo
- N2(midazolam group) (Experimental): Patients in group N2 was treated with intravenous infusion of midazolam on the basis of basic treatment measures which include reducing intracranial pressure with mannitol, hemostasis, acid inhibition, anti-infection, nutrition support and control of blood glucose, blood pressure and body temprature.
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Midazolam — For patients allocated into group N2, 2 mg midazolam will be injected intravenously, and then it will be given at 0.05-0.1 mg/(kg·h) by intravenous infusion. If a surgery is needed, infusion of midazolam will begin 3 hours after the operation and continue for at least 72 hours. During the sedation with midazolam, BIS should be kept at 60 to 80.
  Morphine can be used to supply adequate analgesia.
  Arms: N2(midazolam group)
Drug: Placebo
  Arms: N1(traditional treatment group)

SUMMARY:
To explore the cerebral protective effect of midazolam in patients with traumatic brain injury, we will collect blood samples from patients treated with or without midazolam when the patient is admitted to ICU, 24 h, 48 h and 72 h after the admission before the use of midazolam for patients in group N1, and before the patient is treated with midazolam, 24 h， 48 h, 72 h after the use of midazolam for patients in group N2. Parameters of cerebral metabolism and inflammatory response will be obtained from the blood samples or the cerebrospinal fluid. With the aforementioned parameters, the relationship between clinical outcome and cerebral metabolism and inflammatory response will be detected with statistical method.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or older;
* Hospitalized in ICU within 6 hours after the injury or after the operation;
* Traumatic brain injury is confirmed by computed tomography scan or magnetic resonance imaging, Glasgow Coma Scale is 3 to 12, and the patient should meet the diagnostic standard of severe traumatic brain injury;
* Informed consent is obtained.

Exclusion Criteria:

* Aged less than 18;
* Death is expected in 24 hours;
* History of neurological disease or history of drug abuse which may affect the outcome of the study;
* Failed to obtain Informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Cerebral metabolic parameters | from the admission to ICU to 72 h after the admission for Group N1 and before the use of midazolam to 72 h after the use for group N2
  N1 group: blood samples will be collected when the patient is admitted to ICU, 24 h, 48 h and 72 h after the admission
  N2 group: blood samples will be collected before the use of midazolam, 24 h, 48 h and 72 h after the use
  Blood sample will be collected every time from the radial artery and the jugular bulb separately. The blood sample will be used for blood gas analysis
  Detail parameters by blood test: levels of lactic acid, oxygen saturation(SaO2), partial pressure of oxygen(Pa02), jugular bulb venous oxygen saturation(SjvO2), jugular bulb oxygen partial pressure(PjvO2), hemoglobin(Hb)
  Calculated parameters: arterial oxygen content(Ca02), jugular venous oxygen saturation (SjvO2), arterial venous oxygen content difference(Da-jvO2), cerebral extraction of oxygen(CERO2), Lactate differences between jugular and arterial blood(AVDL) and Cerebral lactate acid production(CLP)
Parameters of intracranial inflammatory response | from the admission to ICU to 72 h after the admission for Group N1 and before the use of midazolam to 72 h after the use for group N2
  N1: blood samples and cerebrospinal fluid are collected when the patient is admitted to ICU, 24 h, 48 h and 72 h after the admission
  N2: blood samples and cerebrospinal fluid are collected before the use of midazolam, 24 h, 48 h and 72 h after the use
  every time, 3 ml blood sample will be collected from the jugular bulb and 2 ml cerebrospinal fluid will be collected at the corresponding time
  The blood sample will be anticoagulated by EDTA and then it will be centrifuged at 3000 r/min for 10 minutes within 30 minutes from the collection. The supernatant liquid will be stored in the freezer at -70℃.
  The cerebrospinal fluid centrifuged at 3000 r/min for 10 minutes, and then the supernatant liquid will be stored in the freezer at -80℃.
  Detail parameters: sFkn and IL-6 levels of the blood sample and CSF will be tested 2 times by ELISA and then take the average.

SECONDARY OUTCOMES:
Ramsay score | from the use of midazolam to 72 h after the use for group N2
seizure | from the admission to ICU to 72 h after the admission
one-week mortality | from the admission to ICU to one week after the admission

CONTACTS AND LOCATIONS:
Locations (1):
- Subei People's Hospital of Jiangsu Province, Yangzhou, Jiangsu, China